CLINICAL TRIAL: NCT04226287
Title: Pilot Study of a Compact Pneumatic Compression Device for Patients With Lymphedema
Brief Title: Compact Pneumatic Compression Device for Patients With Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: A0015
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Lymphedema of Limb

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monterey Pneumatic Compression Device (Experimental): All participants will receive treatment with the Monterey investigational pneumatic compression device
  Interventions: Device: Monterey Pneumatic Compression Device

INTERVENTIONS:
Device: Monterey Pneumatic Compression Device — The MontereyInvestigational System is a compact pneumatic compression device used for the treatment of either primary or secondary lymphedema. The primary intention in this study is to gather usability design feedback. This will be done by observing how a patient uses the device after a brief demonstration from the clinician. Errors and difficulties will be noted by the ResMed representative observing the trial. The qualitative interview with the patient at the end of the trial will yield additional understanding of the patient experience with the device.

SUMMARY:
This is a pilot study for usability and efficacy, and as such it is designed for 15 participants.

The primary objective of this study is to assess the usability of the Monterey Investigational System in the home setting.

The primary objective of this study is to assess the usability of the Monterey Investigational System in the home setting over one week of daily use. Usability will be determined using a 11 point Likert Scale where a score of 10 is considered very favorable and a score of 0 is very unfavorable.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are ≥ 18 years, mentally able to understand and follow the instructions of the study personnel.
* A diagnosis of lower limb Lymphedema.
* Able to provide written and informed consent.
* Patient can read and comprehend English.

Exclusion Criteria:

* Subject undergoing cancer treatment.
* Subject has active lower limb wounds.
* Subject is pregnant or trying to become pregnant.
* History of pulmonary edema or decompensated congestive heart failure.
* Subject has any condition in which increased venous and lymphatic return is undesirable.
* Subject has inbuilt electrical stimulator, e.g., cardiac pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Usability of the Monterey Investigational System in a monitored clinic environment | 1 week
  Usability will be determined using a 11 point Likert Scale where a score of 10 is considered very favorable and a score of 0 is very unfavorable.

SECONDARY OUTCOMES:
Efficacy of Therapy provided by Monterey Investigational system | 1 week
  Efficacy will be determined by comparing lower limb volume measured prior to commencing therapy and at the conclusion. The truncated cone formula is a well-established measure used for assessing limb volume [1]. The limb is divided into segments as per figure 2, measurements taken and volume in each segment is calculated as per the following formula: Voln = L/12(pi)(C1^2+C2^2+C1*C2)

CONTACTS AND LOCATIONS:
Locations (1):
- Progressive Physical Therapy and Rehab, Garden Grove, California, United States

IPD SHARING:
Plan to Share IPD: No